CLINICAL TRIAL: NCT03687359
Title: Prospective, Observational, Longitudinal Study in Pediatric Patients With Moderate to Severe Atopic Dermatitis Whose Disease is Not Adequately Controlled With Topical Prescription Therapies or When Those Therapies Are Not Medically Advisable
Brief Title: Observational Evaluation of Atopic Dermatitis in Pediatric Patients
Acronym: PEDISTAD
Status: Active, not recruiting | Type: Observational
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: OBS15333; U1111-1211-9437 (Registry Identifier: ICTRP)
Record Dates: First submitted 2018-09-06; First posted 2018-09-27 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Dermatitis Atopic
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with atopic dermatitis (AD): Participants receive AD therapy as part of their usual care as determined by their physician independent of decision to enroll in the study.
  Interventions: Other: Standard of care

INTERVENTIONS:
Other: Standard of care — Treatment as per standard practice

SUMMARY:
Primary Objectives:

* To describe the characteristics of pediatric patients with moderate to severe atopic dermatitis (AD) whose disease is not adequately controlled with topical therapies or when those therapies are not medically advisable.
* To evaluate the time-course of AD and selected atopic comorbidities.

Secondary Objectives:

* To characterize disease burden and unmet need.
* To describe real-world treatment patterns (eg, dosing regimens, treatment duration, and reasons for discontinuation and/or switching).
* To document the real-world effectiveness and safety of treatments.

DETAILED DESCRIPTION:
The study duration is 120 months.

ELIGIBILITY:
Inclusion criteria:

* Patients with moderate to severe AD, according to the Investigator's assessment;
* Currently receiving systemic treatment (including phototherapy) for atopic dermatitis or currently on topical treatment, but otherwise candidates for systemic treatment.

Exclusion criteria:

* Concurrent participation in an interventional clinical trial which modifies patient care.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 0 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients with moderate to severe AD whose disease is not adequately controlled with topical therapies or when those therapies are not medically advisable.
Sampling Method: Probability Sample
Enrollment: 1860 (Actual)
Dates: Start 2019-08-15 (Actual); Primary Completion 2035-07-23 (Estimated); Study Completion 2035-07-23 (Estimated)

PRIMARY OUTCOMES:
Patient demographics | Baseline (Month 0)
Medical history of selected atopic diseases and comorbidities | Baseline (Month 0)
Age at onset of atopic dermatitis (AD) | Baseline (Month 0)
Personal and family history of AD and selected atopic diseases | Baseline (Month 0)
All prior and current systemic AD treatment | Baseline (Month 0)
All prior and current topical therapy and phototherapy for AD (including dose, route and frequency of administration for all AD treatment) | Baseline (Month 0)
Presence/severity of AD and selected atopic comorbid conditions | Baseline to Month 120
Therapy for selected atopic comorbid conditions | Baseline to Month 120

SECONDARY OUTCOMES:
Days missed from school for the patient and days missed from work for the primary caregiver due to AD | Baseline to Month 120
Visits to healthcare professionals (HCPs) | Baseline to Month 120
Treatments and prescribing patterns for pediatric AD | Baseline to Month 120
Changes in physician assessment of disease burden (Eczema Area and Severity Index [EASI]) | Baseline to Month 120
Changes in physician assessment of disease burden (Body Surface Area [BSA]) | Baseline to Month 120
Changes in patient/caregiver-reported outcome (PRO): Patient-Oriented Eczema Measure (POEM) | Baseline to Month 120
Change in PRO: Children's Dermatology Life Quality Index (CDLQI)/ Infant's Dermatitis Quality of Life (IDQOL) | Baseline to Month 120
Change in PRO: Dermatitis Family Impact (DFI) | Baseline to Month 120
Change in PRO: Peak Pruritus Numerical Rating Scale (NRS)/ Pruritus (Itch) NRS/ Worst scratching NRS | Baseline to Month 120
Change in PRO: Caregiver Global Assessment of Disease (CGAD) | Baseline to Month 120
Change in PRO: Days missed from school for the patient and days missed from work for the primary caregiver due to AD since last visit | Baseline to Month 120
Change in PRO: Total Nasal Symptom Score (TNSS) | Baseline to Month 120
Change in PRO: Pediatric Asthma Questionnaire (PAQ) | Baseline to Month 120
Change in PRO: Juniper Asthma Control Questionnaire-5 (ACQ-5) | Baseline to Month 120
Adverse event (AE) reporting | Baseline to Month 120

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (182):
- United States (46):
  - C Squared Research Center- Site Number : 8400068, Birmingham, Alabama
  - Cahaba Dermatology & Skin Health Center- Site Number : 8400046, Birmingham, Alabama
  - C2 Research Center, LLC- Site Number : 8400071, Montgomery, Alabama
  - Phoenix Children's Hospital, Inc.- Site Number : 8400015, Phoenix, Arizona
  - Orange County Research Institute- Site Number : 8400028, Anaheim, California
  - Axis Clinical Trials- Site Number : 8400025, Los Angeles, California
  - Madera Family Medical Group- Site Number : 8400054, Madera, California
  - Carey Chronis, MD, FAAP- Site Number : 8400033, Ventura, California
  - Daxia Trials- Site Number : 8400082, Boca Raton, Florida
  - Frieder Dermatology- Site Number : 8400085, Boca Raton, Florida
  - Pediatric Center of Excellence (PCE) - Miami Pediatric Endocrinology, LLC- Site Number : 8400072, Coral Gables, Florida
  - Green Dermatology and Cosmetic Center. Site Number : 8400078, Deerfield Beach, Florida
  - Amedica Research Institute, Inc.- Site Number : 8400067, Hialeah, Florida
  - Eastern Research, Inc.- Site Number : 8400032, Hialeah, Florida
  - Premier Dermatology Partners- Site Number : 8400075, Miami, Florida
  - Nicklaus Children's Hospital - Miami - Southwest 62nd Avenue- Site Number : 8400074, Miami, Florida
  - Vista Health Research, LLC- Site Number : 8400034, Miami, Florida
  - Pediatric & Adult Research Center- Site Number : 8400040, Orlando, Florida
  - Elias Dermatology LLC- Site Number : 8400086, Pembroke Pines, Florida
  - Elias Dermatology LLC- Site Number : 8400087, Pembroke Pines, Florida
  - Centricity Research Talbotton - DBA IACT Health Research at Talbotton Site Number : 8400056, Columbus, Georgia
  - Northwestern University Feinberg School of Medicine- Site Number : 8400001, Chicago, Illinois
  - NorthShore University HealthSystem - Skokie- Site Number : 8400064, Skokie, Illinois
  - The Indiana Clinical Trial Center - Plainfield - Edwards Drive- Site Number : 8400007, Plainfield, Indiana
  - The Indiana Clinical Trials Center, PC Site Number : 8400007, Plainfield, Indiana
  - Michael W. Simon, M.D., PSC- Site Number : 8400073, Lexington, Kentucky
  - Dermatology Associates PC- Site Number : 8400049, Rockville, Maryland
  - Michigan Dermatology Institute Site Number : 8400059, Waterford, Michigan
  - Tokunbo T. Dada, MD PA- Site Number : 8400079, Irvington, New Jersey
  - Family Pediatrics Iwuozo L Obilo Md- Site Number : 8400077, Newark, New Jersey
  - Providence Medical Center- Site Number : 8400081, North Plainfield, New Jersey
  - VAMA Medical Health Center- Site Number : 8400083, Union, New Jersey
  - Park Plaza Dermatology- Site Number : 8400080, New York, New York
  - Philip Fried, M.D., PLLC- Site Number : 8400029, The Bronx, New York
  - Tiga Pediatrics, PC- Site Number : 8400037, The Bronx, New York
  - UNC Hospitals- Site Number : 8400016, Chapel Hill, North Carolina
  - 2G Clinical Research Services- Site Number : 8400031, Durham, North Carolina
  - Clinical Research Of Gastonia- Site Number : 8400041, Gastonia, North Carolina
  - Cincinnati Children's Hospital Medical Center- Site Number : 8400017, Cincinnati, Ohio
  - Dermatology Associates of Mid-Ohio- Site Number : 8400052, Marion, Ohio
  - MUSC- Site Number : 8400013, Charleston, South Carolina
  - ADAC Research- Site Number : 8400048, Greenville, South Carolina
  - Amarillo Center for Clinical Research- Site Number : 8400055, Amarillo, Texas
  - Heights Dermatology & Aesthetic Center- Site Number : 8400065, Houston, Texas
  - The Dermatology Institute of South Texas- Site Number : 8400076, McAllen, Texas
  - Medical College Of Wisconsin- Site Number : 8400008, Milwaukee, Wisconsin
- Argentina (12):
  - Investigational Site Number : 0320009, Bahía Blanca, Buenos Aires
  - Investigational Site Number : 0320003, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Investigational Site Number : 0320004, Rosario, Santa Fe Province
  - Investigational Site Number : 0320007, San Miguel de Tucumán, Tucumán Province
  - Investigational Site Number : 0320006, Buenos Aires
  - Investigational Site Number : 0320001, Buenos Aires
  - Investigational Site Number : 0320002, Buenos Aires
  - Investigational Site Number : 0320008, Buenos Aires
  - Investigational Site Number : 0320005, Ciudad Autonoma Buenos Aires
  - Investigational Site Number : 0320010, Córdoba
  - Investigational Site Number : 0320013, Salta
  - Investigational Site Number : 0320007, San Miguel de Tucumán
- Australia (6):
  - Investigational Site Number : 0360008, Kogarah, New South Wales
  - Investigational Site Number : 0360011, Sydney, New South Wales
  - Investigational Site Number : 0360009, Sydney, New South Wales
  - Investigational Site Number : 0360010, Melbourne, Victoria
  - Investigational Site Number : 0360003, Parkville, Victoria
  - Investigational Site Number : 0360007, Richmond, Victoria
- Brazil (8):
  - Universidade Federal do Paraná- Site Number : 0760003, Curitiba, Paraná
  - Hospital de Clinicas da Universidade Federal do Parana- Site Number : 0760004, Curitiba, Paraná
  - Hospital de Clinicas da Universidade Federal do Parana- Site Number : 0760005, Curitiba, Paraná
  - Irmandade da Santa Casa de Misericórdia de Porto Alegre- Site Number : 0760002, Porto Alegre, Rio Grande do Sul
  - Clinica de Alergia Martti Antila- Site Number : 0760001, Sorocaba, São Paulo
  - IDERJ - Instituto de Dermatologia e Estética do Brasil- Site Number : 0760009, Rio de Janeiro
  - Fundacao Faculdade Regional de Medicina de Sao Jose do Rio Preto- Site Number : 0760007, Sao Jose Rio Preto
  - Hospital Sao Paulo- Site Number : 0760006, São Paulo
- Canada (8):
  - Investigational Site Number : 1240004, Calgary, Alberta
  - Investigational Site Number : 1240007, Calgary, Alberta
  - Investigational Site Number : 1240005, Winnipeg, Manitoba
  - Investigational Site Number : 1240010, Halifax, Nova Scotia
  - Investigational Site Number : 1240001, Markham, Ontario
  - Investigational Site Number : 1240008, Toronto, Ontario
  - Investigational Site Number : 1240006, Montreal, Quebec
  - Investigational Site Number : 1240009, Regina, Saskatchewan
- China (9):
  - Investigational Site Number : 1560004, Beijing
  - Investigational Site Number : 1560006, Changsha
  - Investigational Site Number : 1560001, Chongqing
  - Investigational Site Number : 1560012, Guangzhou
  - Investigational Site Number : 1560007, Harbin
  - Investigational Site Number : 1560005, Shanghai
  - Investigational Site Number : 1560011, Shenzhen
  - Investigational Site Number : 1560002, Suzhou
  - Investigational Site Number : 1560008, Xuzhou
- Colombia (3):
  - Investigational Site Number : 1700006, Barranquilla
  - Investigational Site Number : 1700001, Bogotá
  - Investigational Site Number : 1700004, Bogotá
- Investigational Site Number : 2080002, København NV, Denmark
- France (8):
  - Investigational Site Number : 2500008, Argenteuil
  - Investigational Site Number : 2500001, Bordeaux
  - Investigational Site Number : 2500010, Lille
  - Investigational Site Number : 2500006, Marseille
  - Investigational Site Number : 2500005, Martigues
  - Investigational Site Number : 2500002, Nantes
  - Investigational Site Number : 2500003, Paris
  - Investigational Site Number : 2500011, Toulouse
- Greece (4):
  - Investigational Site Number : 3000004, Larissa
  - Investigational Site Number : 3000005, Thessaloniki
  - Investigational Site Number : 3000003, Thessaloniki
  - Investigational Site Number : 3000002, Thessaloniki
- Israel (5):
  - Investigational Site Number : 3760003, Beersheba
  - Investigational Site Number : 3760004, Haifa
  - Investigational Site Number : 3760005, Kefar Sava
  - Investigational Site Number : 3760001, Ramat Gan
  - Investigational Site Number : 3760002, Rehovot
- Italy (15):
  - Investigational Site Number : 3800004, Terracina, Latina
  - Investigational Site Number : 3800008, Naples, Napoli
  - Investigational Site Number : 3800011, Padua, Padova
  - Investigational Site Number : 3800006, Padua, Veneto
  - Investigational Site Number : 3800012, Bari
  - Investigational Site Number : 3800003, Bologna
  - Investigational Site Number : 3800014, Brescia
  - Investigational Site Number : 3800010, Catania
  - Investigational Site Number : 3800001, Milan
  - Investigational Site Number : 3800005, Napoli
  - Investigational Site Number : 3800015, Pavia
  - Investigational Site Number : 3800009, Perugia
  - Investigational Site Number : 3800013, Reggio Emilia
  - Investigational Site Number : 3800018, Roma
  - Investigational Site Number : 3800007, Trieste
- Japan (18):
  - Investigational Site Number : 3920009, Sagamihara, Kanagawa
  - Investigational Site Number : 3920016, Yokohama, Kanagawa
  - Investigational Site Number : 3920010, Tsu, Mie-ken
  - Investigational Site Number : 3920003, Habikino, Osaka
  - Investigational Site Number : 3920011, Fuchū, Tokyo
  - Investigational Site Number : 3920018, Fukuoka
  - Investigational Site Number : 3920017, Fukuyama-shi
  - Investigational Site Number : 3920002, Hiroshima
  - Investigational Site Number : 3920015, Kumagaya-shi
  - Investigational Site Number : 3920004, Kyoto
  - Investigational Site Number : 3920012, Nagasaki
  - Investigational Site Number : 3920020, Nagoya
  - Investigational Site Number : 3920008, Obu-shi
  - Investigational Site Number : 3920005, Osakasayama-shi
  - Investigational Site Number : 3920014, Sendai
  - Investigational Site Number : 3920019, Sendai
  - Investigational Site Number : 3920001, Tokyo
  - Investigational Site Number : 3920016, Yokohama
- Mexico (8):
  - Investigational Site Number : 4840010, Cuernavaca, Morelos
  - Investigational Site Number : 4840003, Monterrey, Nuevo León
  - Investigational Site Number : 4840009, Monterrey, Nuevo León
  - Investigational Site Number : 4840008, Monterrey, Nuevo León
  - Investigational Site Number : 4840001, México
  - Investigational Site Number : 4840006, México
  - Investigational Site Number : 4840004, Puebla City
  - Investigational Site Number : 4840005, Tlalnepantla
- Netherlands (5):
  - Investigational Site Number : 5280001, Amsterdam
  - Investigational Site Number : 5280005, Groningen
  - Investigational Site Number : 5280002, Rotterdam
  - Investigational Site Number : 5280006, The Hague
  - Investigational Site Number : 5280003, Utrecht
- Norway (3):
  - Investigational Site Number : 5780001, Bergen
  - Investigational Site Number : 5780002, Oslo
  - Investigational Site Number : 5780003, Stavanger
- Portugal (4):
  - Investigational Site Number : 6200003, Braga
  - Investigational Site Number : 6200005, Lisbon
  - Investigational Site Number : 6200001, Lisbon
  - Investigational Site Number : 6200006, Porto
- Russia (5):
  - Investigational Site Number : 6430005, Moscow
  - Investigational Site Number : 6430002, Moscow
  - Investigational Site Number : 6430003, Moscow
  - Investigational Site Number : 6430001, Moscow
  - Investigational Site Number : 6430004, Moscow
- South Korea (7):
  - Investigational Site Number : 4100008, Ansan-si, Gyeonggi-do
  - Investigational Site Number : 4100002, Suwon, Gyeonggi-do
  - Investigational Site Number : 4100007, Incheon, Incheon-gwangyeoksi
  - Investigational Site Number : 4100001, Seoul
  - Investigational Site Number : 4100003, Seoul
  - Investigational Site Number : 4100005, Seoul
  - Investigational Site Number : 4100004, Seoul
- Spain (7):
  - Investigational Site Number : 7240005, Barcelona, Catalunya [Cataluña]
  - Investigational Site Number : 7240012, Pozuelo de Alarcón, Madrid
  - Investigational Site Number : 7240009, Mieres, Principality of Asturias
  - Investigational Site Number : 7240011, Barcelona
  - Investigational Site Number : 7240002, Barcelona
  - Investigational Site Number : 7240003, Madrid
  - Investigational Site Number : 7240010, Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Paller AS, Marcoux D, Ramien M, Baselga E, Carvalho VO, Ardusso LRF, de Graaf M, Pasmans S, Toledo-Bahena M, Rubin C, Joyce JC, Lee LW, Gupta R, Adams B, Ardeleanu M, Zhang A. Systemic Treatments in Moderate-to-Severe Atopic Dermatitis in Pediatric Patients up to 12 Years of Age: Real-World Treatment Outcomes from the PEDISTAD Registry. Am J Clin Dermatol. 2025 Nov;26(6):1031-1043. doi: 10.1007/s40257-025-00962-8. Epub 2025 Sep 19. PMID 40971133
- [Derived] Paller AS, Guttman-Yassky E, Irvine AD, Baselga E, de Bruin-Weller M, Jayawardena S, Zhang A, Mina-Osorio P, Rizova E, Ozturk ZE. Protocol for a prospective, observational, longitudinal study in paediatric patients with moderate-to-severe atopic dermatitis (PEDISTAD): study objectives, design and methodology. BMJ Open. 2020 Mar 24;10(3):e033507. doi: 10.1136/bmjopen-2019-033507. PMID 32209624